CLINICAL TRIAL: NCT00149461
Title: The Efficacy of Written Treatment Plans in Asthma
Brief Title: Written Asthma Actions Plans Versus No Written Instructions In Specialty Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); New York Presbyterian Hospital-Cornell (Unknown); Harlem Hospital Center (Other); Jacobi Medical Center (Other)
Responsible Party: Principal Investigator, David Evans PhD, Professor of Emeritus of Clinical Sociomedical Sciences (In Pediatrics), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA0864; R01HL073955-01 (NIH); R01HL073955 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Asthma Action Plans; African Americans; Latinos; Health Literacy; Asthma Education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Written Asthma Action Plan Group (Experimental): Participants randomized to the written asthma action plan group received an asthma action plan form along with asthma education from their specialist physician.
  Interventions: Behavioral: Written Asthma Action Plan
- No Written Instructions Group (No Intervention): Participants randomized to the usual care group received no written instructions other than prescriptions from their specialist physician.

INTERVENTIONS:
Behavioral: Written Asthma Action Plan
  Other Names: Asthma Treatment Plans; Action Plans
  Arms: Written Asthma Action Plan Group

SUMMARY:
The overall goal of this randomized, controlled study is to compare a model written treatment plan with the usual care that is provided by a group of adult and pediatric pulmonologists and allergists in their practice settings. The written treatment plan is a form that allows a treatment regimen that is consistent with National Heart, Lung, and Blood Institute (NHLBI) guidelines to be conveyed to patients. Barriers to the use of written plans will be identified to better understand why some patients and physicians use written treatment plans more frequently and effectively than others. An additional goal is to assess how patients from different racial/ethnic backgrounds utilize treatments plans. Because asthma disproportionately affects African American and Latino patients, another goal of this study is to better understand if there are fundamental differences in the way patients from racial/ethnic minority groups self-manage asthma in comparison to their white counterparts. The study will also try to determine if differences exist in the way physicians care for minority patients. If there are differences, it is important to determine if the disparities can be overcome with the use of a written treatment plan form.

DETAILED DESCRIPTION:
BACKGROUND:

Effective self-management of asthma requires that patients, or their caregivers, recognize the early symptoms of an exacerbation and initiate appropriate interventions aimed at preventing the progression of symptoms. Most asthma clinical guidelines suggest that the incorporation of a written self-management plan is essential. Patients must possess, understand, and follow a written plan if they are to respond appropriately to changes in asthma status. Nevertheless, there are no controlled studies examining the efficacy of the written plan itself. Furthermore, even if written plans are an essential and effective component of successful self-management, the data suggest that few patients receive these plans. If patients and physicians are to increase their use of written plans, the barriers to the use of these plans need further investigation.

DESIGN NARRATIVE:

The three primary outcome measures of this study are as follows: 1) reduction in asthma symptom frequency; 2) reduction in urgent, unscheduled, and emergency visits for asthma; and 3) improved quality of life. These outcomes will be measured over a 12-month period.

The following four secondary outcome measures will also be examined: 1) hospitalizations due to asthma; 2) days with activity restriction; 3) the proportion of patients in the intervention group who are given the model written plan form during the initial visit; and 4) the proportion of patients in the intervention group who have the model treatment plan at the end of the follow-up period. These outcomes will be measured over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll parents of children (ages 5-17 years) with asthma and adult patients with asthma (ages 18-80 years) who receive care at one of 4 New York Ciry medical centers (New York Presbyterian Hospital-Columbia campus, New York Presbyterian Hospital-Cornell campus, Harlem Hospital Center, and Jacobi Medical Center)
* Diagnosis of persistent asthma (as defined by NHLBI guidelines)
* All participants are new patients to the practice
* Had never been seen by a specialist physician for asthma care
* Had never received a written asthma action plan

Exclusion Criteria:

* Co-morbidity with conditions that affect lung function (e.g, congenital or acquired heart disease, neuromuscular disease, sickle cell disease, or chronic lung disease [bronchopulmonary dysplasia, emphysema, or cystic fibrosis])

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reduction in asthma symptom frequency | Measured at 3 month intervals for 12 months
  Using a 2-week recall period, asthma symptom frequency was measured in 3 ways: (a) the average number of days with asthma symptoms; (b) the average number of nights with symptoms; and (c) the average number of days the participant used a short-acting bronchodilator.
Reduction in urgent, unscheduled, and emergency visits for asthma | Measured at 3 month intervals for 12 months
  Emergency, urgent, and unscheduled visits for asthma were combined into a single measure and assessed using a 3-month recall.
Improved quality of life | Measured at 6 and 12 months
  Asthma QOL, using the Juniper Mini Asthma QOL Scale (MiniAQLQ) for adult participants and the Juniper Pediatric Asthma Caregivers QOL Questionnaire (PACQLQ) for parents, was assessed at 6 and 12-months follow-up.

SECONDARY OUTCOMES:
Hospitalizations due to asthma | Measured at 3 month intervals for 12 months
  Assessed the number of hospital admissions over the previous 3 months.
Days with activity restriction | Measured at 3 month intervals for 12 months
  Days with activity limitations were defined as the number of days missed from school or work due to asthma.
Proportion of participants in the intervention group who are given the written asthma action plan form during the initial visit | Measured at the exit interview after the initial visit with the specialist physician
  Participants in each group show the research assistant all written materials they received from the physician during the visit.
Proportion of patients in the intervention group who have the model treatment plan at the end of the follow-up period | Measured at 12 month interview
  Assessed retention of the written asthma action plan (WAAP) by asking participants to read a specific line from the written asthma action plan to demonstrate that they had the WAAP in their possession.

CONTACTS AND LOCATIONS:
Overall Officials: David Evans, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Result] Sheares BJ, Du Y, Vazquez TL, Mellins RB, Evans D. Use of written treatment plans for asthma by specialist physicians. Pediatr Pulmonol. 2007 Apr;42(4):348-56. doi: 10.1002/ppul.20586. PMID 17352397
- [Derived] Sheares BJ, Mellins RB, Dimango E, Serebrisky D, Zhang Y, Bye MR, Dovey ME, Nachman S, Hutchinson V, Evans D. Do Patients of Subspecialist Physicians Benefit from Written Asthma Action Plans? Am J Respir Crit Care Med. 2015 Jun 15;191(12):1374-83. doi: 10.1164/rccm.201407-1338OC. PMID 25867075